CLINICAL TRIAL: NCT00317421
Title: Effects of Regular Treatment With Sildenafil on Blood Pressure and Endothelial Function in Untreated Hypertensives
Brief Title: Effect of Regular Sildenafil on Blood Pressure and Arterial Function in Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: JO-02
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Last update posted 2006-04-24 (Estimated); Status verified 2004-02

CONDITIONS: Hypertension
Keywords: Phosphodiesterase 5; Sildenafil; Hypertension; Blood pressure; Arterial stiffness; Endothelial function
MeSH Terms: conditions — Hypertension | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: Sildenafil citrate

SUMMARY:
The purpose of the study is to investigate if regular treatment with sildenafil reduces blood pressure and improves blood vessel function in patients with hypertension (high blood pressure).

DETAILED DESCRIPTION:
Inhibitors of phosphodiesterase type 5 (PDE5), such as sildenafil, relax blood vessels. In the penis this facilitates erection and sildenafil has proved a very effective treatment for male erectile dysfunction.

To date, most work on the effects of sildenafil on blood pressure have mainly been investigated in single dose studies. These have shown that sildenafil causes a modest reduction in blood pressure, even when taken with other blood pressure-lowering drugs, providing reassurance on safety when taken as a single dose for erectile dysfunction. However, these studies do not offer any insight into the potential of PDE5 inhibition in the long-term treatment of hypertension. We will address this question by investigating the effects of regular administration of sildenafil on blood pressure. It may also be postulated that, because of its mechanism of action, sildenafil will also improve the function of the endothelium, the single layer of cells that lines all blood vessels. Therefore, the effect of regular sildenafil on endothelial function in hypertension will also be investigated in the study.

The study will be performed in a randomised, placebo-controlled, double blind, 2-way crossover manner. Sildenafil and matched placebo will each will taken three times daily for 2 weeks, with a washout of at least 6 days between treatments. Measurements will be made acutely (before and 1 hour after oral sildenafil) of heart rate, blood pressure, pulse wave analysis (a measure of wave reflection in arteries), pulse wave velocity (a measure of arterial stiffness) and flow-mediated dilatation (a measure of endothelial function). These measurements will be repeated 2 weeks later (again just before and 1 hour after oral sildenafil). In addition, ambulatory blood pressure will be recorded after 2 weeks of treatment (baseline ambulatory BP will be taken as the recording made at diagnosis).

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Hypertensive (office systolic BP ≥160 mmHg or diastolic BP ≥100 mmHg), not taking antihypertensive drugs OR hypertensive controlled (systolic BP < 160 mmHg or diastolic BP < 100 mmHg) on 1 antihypertensive agent
* Hypertension confirmed on ambulatory monitoring (average daytime BP ≥145/95 mmHg)
* Patients will also be included if they have 'borderline' hypertension and their calculated 10-year risk of cardiovascular disease is >20% or they have target organ damage. Borderline hypertension will be defined according to ambulatory BP criteria alone (average awake systolic BP ≥135 and <145 mmHg or diastolic BP ≥85 and <95 mmHg).

Exclusion Criteria:

* History of other major cardiac, respiratory, neurological or renal disease
* Systolic BP consistently >210 mmHg or diastolic BP consistently >120 mmHg
* Systolic BP consistently >180 mmHg or diastolic BP consistently >110 mmHg in those withdrawn from existing therapy
* Current alcohol abuse
* Diabetes
* Taking vasoactive drugs
* Previous serious drug allergy
* Pregnant
* Participation, within 6 months, in other research studies

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2004-03; Study Completion 2005-11

PRIMARY OUTCOMES:
Change in blood pressure
Change in flow-mediated dilatation
Change in central augmentation index (derived from pulse wave analysis)
Change in carotid-femoral pulse wave velocity

CONTACTS AND LOCATIONS:
Overall Officials: James J Oliver, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Clinical Pharmacology Unit, University of Edinburgh, Edinburgh, Lothian, United Kingdom

REFERENCES:
- [Background] Zusman RM, Morales A, Glasser DB, Osterloh IH. Overall cardiovascular profile of sildenafil citrate. Am J Cardiol. 1999 Mar 4;83(5A):35C-44C. doi: 10.1016/s0002-9149(99)00046-6. PMID 10078541